CLINICAL TRIAL: NCT02287714
Title: Surgical Treatment of Plantar Fasciitis: Instep Plantar Fasciotomy With and Without Gastrocnemius Recession
Brief Title: Instep Plantar Fasciotomy With and Without Gastrocnemius Recession
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low (no) enrollment.
Sponsor: OhioHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0043
Record Dates: First submitted 2014-10-07; First posted 2014-11-11 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Plantar Fasciitis; Equinus Deformity
Keywords: Instep plantar fasciotomy
MeSH Terms: conditions — Fasciitis, Plantar; Equinus Deformity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Instep without Gastrocnemius Recession (Active Comparator): Patient will receive an instep plantar fascial release but not a gastrocnemius recession.
  Interventions: Procedure: Instep without gastrocnemius recession
- Instep with Gastrocnemius Recession (Experimental): Patient will receive an instep plantar fascial release as well as a gastrocnemius recession.
  Interventions: Procedure: Instep with gastrocnemius recession

INTERVENTIONS:
Procedure: Instep without gastrocnemius recession — Patient will receive an instep plantar fascial release without gastrocnemius recession.
  Arms: Instep without Gastrocnemius Recession
Procedure: Instep with gastrocnemius recession — Patient will receive an instep plantar fascial release as well as gastrocnemius recession.
  Arms: Instep with Gastrocnemius Recession

SUMMARY:
Compare results of Instep Plantar Fascial release with and without gastrocnemius recession

DETAILED DESCRIPTION:
Plantar fasciitis is one of the most common causes of heel pain. Approximately 2 million Americans seek treatment for plantar fasciitis every year, with 10% of the population developing plantar fasciitis over a lifetime. The vast majority of cases respond to conservative care; however, the 5-10% of cases that are recalcitrant to conservative measures may require surgical intervention. Several surgical options do exist and are cited in the literature for treatment of recalcitrant plantar fasciitis. One such approach is the instep plantar fascial release, utilizing an approximately 2-3 cm plantar incision over the prominent fascial band, just distal to the fat pad of the heel. It has been demonstrated that many patients with plantar fasciitis also have an isolated contracture of the gastrocnemius, known as gastrocnemius equinus. Gastrocnemius recession is performed to correct an isolated gastrocnemius contracture and recent studies have demonstrated its successful use in the treatment of recalcitrant foot pain. To date, no prospective studies exist examining the utilization of the gastrocnemius recession in combination with instep plantar fascial release in the treatment of recalcitrant plantar fasciitis. This prospective randomized trial will aim to compare the use of instep plantar fasciotomy both with and without gastrocnemius recession in the treatment of plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have failed conservative treatment for greater than 6 months.
* Patients with recalcitrant plantar fasciitis and simultaneous gastrocnemius contracture in the ipsilateral limb. Contracture will be defined as the inability to dorsiflex the ankle past neutral with the knee in extension.

Exclusion Criteria:

* Adjunctive procedure at the time of surgery.
* History of heel spur surgery, plantar fasciotomy or extracorporeal shockwave therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in American Orthopedic Foot and Ankle Society Score | change from baseline (within 30 days prior to intervention) AOFAS score at 3 mo, 6 mo, and one year
  Subjective and objective measurements which scale a patients' pain and function collected at selected intervals and compared to pre-operatively.

SECONDARY OUTCOMES:
Adjunctive treatment | One year
  Participant chart will be reviewed for any adjunctive treatment required following their surgical intervention
Complications | One year
  Participant chart will be reviewed for any complications that occurred during their one year follow-up, including but not limited to: Recurrence of symptoms, no improvement, infection, tear or rupture of plantar fascia following procedure
Change in Activity level | change from baseline (within 30 days prior to intervention) activity level at 3 months, 6 months, and one year
  A patient submitted survey regarding their activity level and ability to perform those activities pain free.
Change Pain level | change from baseline (within 30 days prior to intervention) pain level at 3 months, 6 months, and one year
  Patients will be asked to submit their pain level utilizing the Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Quisno, DPM, Principal Investigator — OhioHealth
Locations (4):
- United States (4):
  - Step Lively Foot and Ankle Center, Dublin, Ohio
  - Foot and Ankle Specialists of Central Ohio, Gahanna, Ohio
  - Step Lively Foot and Ankle Center, Grove City, Ohio
  - Step Lively Foot and Ankle Center, Reynoldsburg, Ohio